CLINICAL TRIAL: NCT07334535
Title: A Prospective, Randomized, Multi-center Study Comparing Isatuximab in Combination With VRD Versus VRD in High-Risk, Transplant-Ineligible Patients With Newly Diagnosed Multiple Myeloma.
Brief Title: Isa-VRD in TIE HRMM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Handan Central Hospital (Other); Inner Mongolia People's Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Hebei Medical University Third Hospital (Other); North China University of Science and Technology (Other); China-Japan Union Hospital, Jilin University (Other); Cangzhou Central Hospital (Other); Yantai Yuhuangding Hospital (Other); Shengjing Hospital (Other); Second Hospital of Shanxi Medical University (Other); Beijing Chao Yang Hospital (Other); Beijing Jishuitan Hospital (Other); Henan Cancer Hospital (Other Government); Beijing Hospital (Other Government); Xuanwu Hospital, Beijing (Other); Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Junling Zhuang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K9520; 2025-PUMCH-C-040 (Other Grant/Funding Number: National High Level Hospital Clinical Research)
Record Dates: First submitted 2026-01-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; isatuximab; RCT
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IsaVRD group (Experimental): Participants in this group will receive the quadruplet induction-consolidation regimen of Isatuximab in combination with Bortezomib, Lenalidomide, and Dexamethasone (Isa-VRD) for 12 cycles (each cycle is 28 days). This will be followed by a maintenance therapy with Isatuximab, Bortezomib and Lenalidomide until disease progression or unacceptable toxicity.
  Interventions: Drug: Isatuximab, bortezomib, lenalidomide, dexamethason
- VRD group (Active Comparator): Participants in this group will receive the standard triplet induction-consolidation regimen of Bortezomib, Lenalidomide, and Dexamethasone (VRD) for 12 cycles (each cycle is 28 days). This will be followed by a maintenance therapy with Bortezomib and Lenalidomide until disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib, Lenalidomide, Dexamethasone

INTERVENTIONS:
Drug: Isatuximab, bortezomib, lenalidomide, dexamethason — Participants in this group will receive the quadruplet induction-consolidation regimen of Isatuximab in combination with Bortezomib, Lenalidomide, and Dexamethasone (Isa-VRD) for 12 cycles (each cycle is 28 days). This will be followed by a maintenance therapy with Isatuximab, Bortezomib and Lenalidomide until disease progression or unacceptable toxicity.
  Arms: IsaVRD group
Drug: Bortezomib, Lenalidomide, Dexamethasone — Participants in this group will receive the standard triplet induction-consolidation regimen of Bortezomib, Lenalidomide, and Dexamethasone (VRD) for 12 cycles (each cycle is 28 days). This will be followed by a maintenance therapy with Bortezomib and Lenalidomide until disease progression or unacceptable toxicity.
  Arms: VRD group

SUMMARY:
This is a multicenter, prospective, randomized controlled trial designed to compare the quadruplet regimen of isatuximab, bortezomib, lenalidomide, and dexamethasone (Isa-VRD) with the standard triplet regimen (VRD) in newly diagnosed, transplant-ineligible patients with high-risk multiple myeloma (HRMM).

Primary Hypothesis:

The addition of isatuximab to VRD will significantly improve the MRD negativity rate at 12 months compared to VRD alone in HR-NDMM patients.

Secondary Hypotheses:

Isa-VRD will lead to higher overall response rates (ORR), deeper responses, and improved progression-free survival (PFS) and overall survival (OS).

The safety profile of Isa-VRD will be manageable and consistent with the known safety profiles of its individual components.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, open-label, Phase IIIb clinical trial. The study aims to evaluate the efficacy and safety of the quadruplet regimen Isatuximab in combination with Bortezomib, Lenalidomide, and Dexamethasone (Isa-VRD) compared to the standard triplet regimen of Bortezomib, Lenalidomide, and Dexamethasone (VRD) in newly diagnosed high-risk multiple myeloma (HRMM) patients who are not candidates for autologous stem cell transplantation.

A total of 117 participants will be enrolled and randomly assigned in a 2:1 ratio to receive either Isa-VRD (78 participants) or VRD (39 participants). The study consists of an induction-consolidation phase (cycles 1-12) followed by a maintenance phase (from cycle 13 onwards until disease progression or unacceptable toxicity).

The primary endpoint is the rate of minimal residual disease (MRD) negativity in the bone marrow assessed by flow cytometry at 12 months of treatment. Key secondary endpoints include MRD negativity rate at 18 months, objective response rate (ORR), progression-free survival (PFS), overall survival (OS), and safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Multiple myeloma ，meeting the IMWG 2025 definition of high-risk MM (any one criterion):

  (1) Del(17p) (>20% of plasma cells) and/orTP53 mutation or（2）One of these translocations cooccurring with 1q+ and/or del(1p32) , or t(4;14), or t(14;16), or t(14;20) or （3） Monoallelic del(1p32) along with 1q+ or biallelic del(1p32) or（4） High β2M (>5.5 mg/dL) with normal creatinine (<1.2 mg/dL) or（5）Or presents with any other high-risk feature: meeting diagnostic criteria for primary plasma cell leukemia or presence of extramedullary plasmacytoma at baseline;
* Age ≥18 years and ≤80 years;
* Not eligible for autologous hematopoietic stem cell transplantation or has declined transplantation for other reasons.
* ECOG score 0-2
* Expected survival time > 3 months
* Sufficient organ function is defined as follows: absolute neutrophil count ≥ 1.0×10^9/L, platelet count ≥ 50×10^9/L (when the proportion of bone marrow plasma cells is <50%), hemoglobin ≥ 7.5 g/dL; total bilirubin ≤ 1.5 times the upper limit of normal, aspartate aminotransferase and alanine aminotransferase ≤ 2.5 times the upper limit of normal; creatinine clearance rate ≥ 30 mL/min; left ventricular ejection fraction ≥ 50%.
* Fertile female or male subjects must agree to take effective contraceptive measures during the study period and within the specified time after the last administration.
* Voluntarily participated in this study, signed the informed consent form, had good compliance, and was cooperative during the follow-up.

Exclusion Criteria:

* Prior systemic anti-myeloma therapy;
* Viral infections including HBV, HCV, HIV, etc.;
* Serious cardiovascular and cerebrovascular diseases, such as: within 6 months before screening, myocardial infarction, unstable angina pectoris, severe arrhythmia, New York Heart Function Classification III-IV grade, or left ventricular ejection fraction <50%.
* Severe neurological or mental disorders that affect the ability to give informed consent or comply with the protocol.
* Had an allergic reaction to isatuximab, bortezomib, lenalidomide, dexamethasone or any excipients
* Pregnant or lactating women.
* Participated in other interventional clinical studies, or had received other anti-tumor treatments within the specified time before the first administration of this study.
* The researcher believes that there are any other circumstances unsuitable for participating in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
MRD negativity rate at 12 months | at 12 months post-treatment initiation
  MRD negativity rate at 12 months post-treatment initiation, assessed by EuroFlow (NGF) with a sensitivity of at least 10-5

SECONDARY OUTCOMES:
MRD negativity rate at 18 months | at 18 months post-treatment initiation
  MRD negativity rate at 18 months post-treatment initiation, assessed by EuroFlow (NGF) with a sensitivity of at least 10-5
Progression-free survival | From date of enrollment until the date of first documented progression
  from enrollment to first disease progression
overall survival | : From date of enrollment until the date of death from any cause
  from enrollment to death with follow-up
Overall response rate | From randomization until the end of the induction-consolidation phase
  The proportion of participants who achieve a predefined response or better according to the International Myeloma Working Group (IMWG) uniform response criteria. The response categories included in the ORR calculation are: stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), and Partial Response (PR). ORR will be calculated as (number of participants with sCR+CR+VGPR+PR) / (total number of response-evaluable participants) * 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Junling Zhuang, Study Chair — Peking Union Medical College, department of hematology
Locations (1):
- Junling Zhuang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
individual baseline characteristic, treatment and follow-up results will be shared after publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication, the data will become available

REFERENCES:
- [Background] Davies FE, Pawlyn C, Usmani SZ, San-Miguel JF, Einsele H, Boyle EM, Corre J, Auclair D, Cho HJ, Lonial S, Sonneveld P, Stewart AK, Bergsagel PL, Kaiser MF, Weisel K, Keats JJ, Mikhael JR, Morgan KE, Ghobrial IM, Orlowski RZ, Landgren CO, Gay F, Caers J, Chng WJ, Chari A, Walker BA, Kumar SK, Costa LJ, Anderson KC, Morgan GJ. Perspectives on the Risk-Stratified Treatment of Multiple Myeloma. Blood Cancer Discov. 2022 Jul 6;3(4):273-284. doi: 10.1158/2643-3230.BCD-21-0205. PMID 35653112
- [Background] Facon T, Dimopoulos MA, Leleu XP, Beksac M, Pour L, Hajek R, Liu Z, Minarik J, Moreau P, Romejko-Jarosinska J, Spicka I, Vorobyev VI, Besemer B, Ishida T, Janowski W, Kalayoglu-Besisik S, Parmar G, Robak P, Zamagni E, Goldschmidt H, Martin TG, Manier S, Mohty M, Oprea C, Bregeault MF, Mace S, Berthou C, Bregman D, Klippel Z, Orlowski RZ; IMROZ Study Group. Isatuximab, Bortezomib, Lenalidomide, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2024 Oct 31;391(17):1597-1609. doi: 10.1056/NEJMoa2400712. Epub 2024 Jun 3. PMID 38832972
- [Background] Leleu X, Hulin C, Lambert J, Bobin A, Perrot A, Karlin L, Roussel M, Montes L, Cherel B, Chalopin T, Slama B, Chretien ML, Laribi K, Dingremont C, Roul C, Mariette C, Rigaudeau S, Calmettes C, Dib M, Tiab M, Vincent L, Delaunay J, Santagostino A, Macro M, Bourgeois E, Orsini-Piocelle F, Gay J, Bareau B, Bigot N, Vergez F, Lebreton P, Tabrizi R, Waultier-Rascalou A, Frenzel L, Le Calloch R, Chalayer E, Braun T, Lachenal F, Corm S, Kennel C, Belkhir R, Blade JS, Joly B, Richez-Olivier V, Gardeney H, Demarquette H, Robu-Cretu D, Garderet L, Newinger-Porte M, Kasmi A, Royer B, Decaux O, Arnulf B, Belhadj K, Touzeau C, Mohty M, Manier S, Moreau P, Avet-Loiseau H, Corre J, Facon T. Isatuximab, lenalidomide, dexamethasone and bortezomib in transplant-ineligible multiple myeloma: the randomized phase 3 BENEFIT trial. Nat Med. 2024 Aug;30(8):2235-2241. doi: 10.1038/s41591-024-03050-2. Epub 2024 Jun 3. PMID 38830994
- [Background] Deckert J, Wetzel MC, Bartle LM, Skaletskaya A, Goldmacher VS, Vallee F, Zhou-Liu Q, Ferrari P, Pouzieux S, Lahoute C, Dumontet C, Plesa A, Chiron M, Lejeune P, Chittenden T, Park PU, Blanc V. SAR650984, a novel humanized CD38-targeting antibody, demonstrates potent antitumor activity in models of multiple myeloma and other CD38+ hematologic malignancies. Clin Cancer Res. 2014 Sep 1;20(17):4574-83. doi: 10.1158/1078-0432.CCR-14-0695. Epub 2014 Jul 1. PMID 24987056